CLINICAL TRIAL: NCT01725828
Title: Ultrasound is Superior to Conventional Palpation Method in Identification of the Cricothyroid Membrane in Subjects With Poorly Defined Neck Landmarks: A Randomized Clinical Trial
Brief Title: Accuracy of Ultrasound in Identification of Cricothyroid Membrane: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Principal Investigator, Dr. Naveed Siddiqui, Associate Professor, Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1-2012
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Difficult Breathing
Keywords: Cricothyroid membrane; Ultrasound; Neck landmarks; External palpation
MeSH Terms: conditions — Dyspnea | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- External Palpation group (Experimental): External Palpation group will consist of 109 patients, who's CTM will be marked using traditional palpation technique of identifying the Cricothyroid membrane.
  Interventions: Other: External Palpation
- Ultrasound group (Experimental): Ultrasound group will consist of 114 patients, who's CTM will be marked using, ultrasonography to identify the CTM.
  The Intervention by using the Ultrasound to determine the CTM.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Using the Ultrasound to determine the location of the CTM.
  Other Names: Ultrasonography
  Arms: Ultrasound group
Other: External Palpation — Using External Palpation to identify cricothyoid membrane
  Other Names: Digital Palpation
  Arms: External Palpation group

SUMMARY:
Routine surgery requires artificial breathing through the placement of a plastic tube into the patient's windpipe via mouth or nose. This tube serves as the source of providing oxygen to the patients during surgery. Difficulties during insertion of this tube may lead to serious complications and during this life-threatening crisis the only way to provide oxygen to the patient is by the help of a procedure called cricothyrotomy (CTY).

CTY is a life saving procedure that involves an incision on the patient neck at a very precise location called Cricothyroid Membrane (CTM). The current method of identifying this location is by palpation of neck cartilages by the operator. The incorrect identification of the CTM could lead to many complications. In certain patients such as obese or distorted neck features the identification of CTM would be difficult. Ultrasound (US) has improved the success rate of many anesthesia procedures .Its use has been described for identification of neck structures; however, this technique of localization has not been validated against the gold standard which is the use of CT scan. The purpose of our study is to determine the precision of identifying the CTM using the US versus the conventional finger palpation when compared to the gold standard.

DETAILED DESCRIPTION:
Inability to secure the airway remains the most frequent cause of anesthesia-related mishaps.Difficult airway management continues to be the major challenge in anesthesia as it is responsible for a third of anesthesia-related claims and is the single largest class of closed claim injury suits. Difficulties in tracheal intubation is the most frequent cause of anesthesia-related morbidity and mortality.

Repeated attempts of tracheal intubations can result in serious soft tissue injury and rapidly deteriorate into a life threatening "cannot intubate-cannot ventilate" (CICV) crisis. The guidelines suggested by the American Society of Anesthesiologists and the Difficult Airway Society for managing the unanticipated difficult airway recommend the performance of a cricothyrotomy(CTY) as the next step for a CICV scenario.

Cricothyrotomy is an infrequently performed life saving procedure when facing a difficult CICV airway.Previous studies quote, the incidence of the CICV scenario to be in the range of 0.01-2 per 10,000 cases. It is therefore imperative that anesthesiologists have the necessary knowledge and skills in successfully managing this life-threatening airway crisis. However, several studies demonstrated that many practicing anesthesiologists and anesthesia trainees (residents/fellows) are uncomfortable with the management of a CICV situation because it is such a rare event. A recent Canadian survey shows that only a quarter of the residents and 40% of practicing anesthesiologists were comfortable with performing a cricothyrotomy. Similar findings were reported in a German national survey of academic teaching hospitals where difficult airway situations, particularly a CICV crisis, were poorly managed and were postulated to have contributed to adverse patient outcomes.Complications of emergency CTY by physicians are common, with rates ranging from 9% to 40%.These complications include failure to cannulate the trachea, false airway passage, severe bleeding, posterior tracheal wall injuries, pneumothorax and esophageal laceration. All of these major complications may be related to improper identification of anatomical landmarks used to identify the correct position of cricothyroid membrane (CTM). The current method of CTY relies solely on digital palpation of these landmarks to accurately identify the CTM.

Several studies have identified independent predictors for patients with difficult airway. These include characteristics such as high body mass index, presence of beard, short bull neck, distorted neck anatomy either due to congenital or acquired pathology such as goiters or radiation to the neck. These are the same factors which may lead to improper identification of neck landmarks for the CTY.

The outcome and accuracy of CTY may be improved with better preparedness and pre-procedural identification of the neck landmarks for CTY before deciding the method of anesthetic. This is especially true in patients with anatomical features of difficult airway, who may be the ones more likely to have a difficult airway or require an emergency CT. In this patient population, incorrect localization of the CTM may lead to significant airway morbidity or failure to quickly establish an airway.

The role of ultrasound in airway management:

Bedside ultrasound is increasingly being used to assist anesthesiologists in performing various procedures.The use of ultrasonography (US) has been shown to significantly reduce complications and improve outcomes. Diagnostic application of US for upper airway anatomy and its role for the performance of CTY and bedside tracheostomy has been previously described. However, little is known on the reliability and validity of the US when compared to the gold standard CT scan in identifying the CTM.

The methods used to identify CTM are based on identification of anatomical landmarks and digital palpation. This may be difficult in patients with poorly defined anatomy, the very same population in which the likelihood of a difficult intubation/emergency surgical airway are higher.

The trachea and paratracheal soft tissues of the neck can be examined at the highest resolution with US probes of high frequency due to their superﬁcial position. The anterior tracheal wall, thyroid and cricoid cartilages, tracheal rings, and pre-tracheal tissue may all be well visualized , which allows the clinician to select the optimal space for CTY tube placement. The use of US for assisting with airway management in anesthesia and in the intensive care unit is directly related to the availability of low-cost and portable US capabilities. Clinicians initially described US-guided central venous catheterization, followed by US-guided regional anesthesia techniques. Recently, a few studies examined the role of US for emergency airway procedures. Nichollas et al developed a standardized US technique to identify the CTM. The findings in this study suggest that the CTM and relevant structures can be quickly identified by emergency physicians using US technique. However this study was limited to patients with normal airway and mainly focused to the standardization of technique. it did not validate the technique against a gold standard. In another study Muhammad et al, reported four cases in which ultrasound was successfully used to perform percutaneous tracheostomy in the ICU. Cricothyroid membrane can easily be located on CT scan.

In summary, inability to secure the airway remains the most frequent cause of anesthesia-related morbidity and mortality. CTY is highly dependent on proper identification of anatomical land-marks.

ELIGIBILITY:
Inclusion Criteria:

ASA physical status I-III patients aged ≥ 18 with neck pathology who were scheduled for a neck CT scan at University Health Network. All patients recruited in the study had neck pathologies including previous neck surgery, irradiation and/or neck mass.

Exclusion Criteria:

patients who were unable to lie flat, unable to maintain a neutral neck position and those who refused to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
accuracy in identification of the Cricothyroid Membrane | Less than 1 min
  accuracy in identification of the CM which was measured by a digital ruler in millimeter from the CT-point to the US-point or EP-point. We defined success as the proportion of accurate attempts within 5 mm distance from the CT-point to the US-point or EP-point.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Siddiqui, MD, MSc, Principal Investigator — Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Locations (2):
- Canada (2):
  - UHN, Toronto, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Result] Caplan RA, Posner KL, Ward RJ, Cheney FW. Adverse respiratory events in anesthesia: a closed claims analysis. Anesthesiology. 1990 May;72(5):828-33. doi: 10.1097/00000542-199005000-00010. PMID 2339799
- [Result] Domino KB, Posner KL, Caplan RA, Cheney FW. Airway injury during anesthesia: a closed claims analysis. Anesthesiology. 1999 Dec;91(6):1703-11. doi: 10.1097/00000542-199912000-00023. PMID 10598613
- [Result] American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Practice guidelines for management of the difficult airway: an updated report by the American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Anesthesiology. 2003 May;98(5):1269-77. doi: 10.1097/00000542-200305000-00032. No abstract available. PMID 12717151
- [Result] Segal R. A response to 'Difficult Airway Society guidelines for management of the unanticipated difficult intubation', Henderson JJ, Popat MT, Latto IP and Pearce AC, Anaesthesia 2004; 59: 675-94. Anaesthesia. 2004 Nov;59(11):1150-1. doi: 10.1111/j.1365-2044.2004.04005.x. No abstract available. PMID 15479346
- [Result] Mori M, Fujimoto J, Iwasaka H, Noguchi T. Emergency percutaneous dilatational cricothyroidotomy after failed intubation. Anaesth Intensive Care. 2002 Feb;30(1):101-2. No abstract available. PMID 11939430
- [Result] Griggs WM, Myburgh JA, Worthley LI. Urgent airway access--an indication for percutaneous tracheostomy? Anaesth Intensive Care. 1991 Nov;19(4):586-7. doi: 10.1177/0310057X9101900421. No abstract available. PMID 1750647
- [Result] Goldmann K, Braun U. Airway management practices at German university and university-affiliated teaching hospitals--equipment, techniques and training: results of a nationwide survey. Acta Anaesthesiol Scand. 2006 Mar;50(3):298-305. doi: 10.1111/j.1399-6576.2006.00853.x. PMID 16480462
- [Result] Wong DT, Lai K, Chung FF, Ho RY. Cannot intubate-cannot ventilate and difficult intubation strategies: results of a Canadian national survey. Anesth Analg. 2005 May;100(5):1439-1446. doi: 10.1213/01.ANE.0000148695.37190.34. PMID 15845702
- [Result] Bair AE, Panacek EA, Wisner DH, Bales R, Sakles JC. Cricothyrotomy: a 5-year experience at one institution. J Emerg Med. 2003 Feb;24(2):151-6. doi: 10.1016/s0736-4679(02)00715-1. PMID 12609644
- [Result] McGill J, Clinton JE, Ruiz E. Cricothyrotomy in the emergency department. Ann Emerg Med. 1982 Jul;11(7):361-4. doi: 10.1016/s0196-0644(82)80362-4. PMID 7091796
- [Result] Hsiao J, Pacheco-Fowler V. Videos in clinical medicine. Cricothyroidotomy. N Engl J Med. 2008 May 29;358(22):e25. doi: 10.1056/NEJMvcm0706755. No abstract available. PMID 18509116
- [Result] Kumar A, Chuan A. Ultrasound guided vascular access: efficacy and safety. Best Pract Res Clin Anaesthesiol. 2009 Sep;23(3):299-311. doi: 10.1016/j.bpa.2009.02.006. PMID 19862889
- [Result] Levin PD, Sheinin O, Gozal Y. Use of ultrasound guidance in the insertion of radial artery catheters. Crit Care Med. 2003 Feb;31(2):481-4. doi: 10.1097/01.CCM.0000050452.17304.2F. PMID 12576955
- [Result] Warman P, Nicholls B. Ultrasound-guided nerve blocks: efficacy and safety. Best Pract Res Clin Anaesthesiol. 2009 Sep;23(3):313-26. doi: 10.1016/j.bpa.2009.02.004. PMID 19862890
- [Result] Erkan M, Tolu I, Aslan T, Guney E. Ultrasonography in laryngeal cancers. J Laryngol Otol. 1993 Jan;107(1):65-8. doi: 10.1017/s0022215100122182. PMID 8445322
- [Result] Sustic A, Zupan Z, Antoncic I. Ultrasound-guided percutaneous dilatational tracheostomy with laryngeal mask airway control in a morbidly obese patient. J Clin Anesth. 2004 Mar;16(2):121-3. doi: 10.1016/j.jclinane.2003.04.005. PMID 15110374
- [Result] Muhammad JK, Patton DW, Evans RM, Major E. Percutaneous dilatational tracheostomy under ultrasound guidance. Br J Oral Maxillofac Surg. 1999 Aug;37(4):309-11. doi: 10.1054/bjom.1999.0072. PMID 10475654
- [Result] Nicholls SE, Sweeney TW, Ferre RM, Strout TD. Bedside sonography by emergency physicians for the rapid identification of landmarks relevant to cricothyrotomy. Am J Emerg Med. 2008 Oct;26(8):852-6. doi: 10.1016/j.ajem.2007.11.022. PMID 18926340
- See also: Cricothyroidotomy is indicated upon failure to obtain an airway — http://emedicine.medscape.com/article/1830008-overview
- See also: Ultrasound Assisted Cricothyrotomy — http://www.youtube.com/watch?v=z0egxtce0LQ
- See also: Ultrasound Guided Versus Palpation Guided Cricothyrotomy With Poorly Defined Anatomical Landmarks — http://clinicaltrials.gov/ct2/show/NCT01475487